CLINICAL TRIAL: NCT04874077
Title: Using Voice Biomarkers to Predict the Likelihood of Major Depressive Disorder: A Multi-Site Fully Remote E-Clinical Validation Study
Brief Title: Using Voice Biomarkers to Predict the Likelihood of Major Depressive Disorder
Status: Completed | Type: Observational
Sponsor: Kintsugi Mindful Wellness, Inc. (Industry)
Collaborators: San Francisco Psychiatry Group (Unknown); Frontier Psychiatry (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2021/03/20
Record Dates: First submitted 2021-04-30; First posted 2021-05-05 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-06

CONDITIONS: Major Depressive Disorder
Keywords: Voice biomarkers; Speech analysis
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Case
- Control

SUMMARY:
Major Depressive Disorder (MDD) is the leading cause of disability worldwide. Depression and anxiety disorders are among the most prevalent of all mental disorders, with an estimated annual prevalence of 9.7% and 18.1% respectively.

It has been known for the last 100 years that depression and anxiety both likely affect vocal acoustic properties. In 1921, Emil Kraepelin, characterized depressed patient's voices as having a lower pitch, lower volume, lower rate of speech, more monotony of prosody as well as more hesitations, stuttering, and whispering.

Mechanistically, it is possible that the neural circuitry involved in the pathophysiology of mood and anxiety disorders impinge upon the neural circuit involved in speech production, affecting qualities that include rate, prosody, speech latency and other paralinguistic features. Thus, acoustic features of speech may be one of the more readily accessible biomarkers for these conditions.

Given this understanding, the investigators sought to develop a passive vocal biomarker instrument for depression and anxiety screening that could markedly expand access as well as standardize the quality of screening in primary care settings.

ELIGIBILITY:
Inclusion Criteria:

* Adult males and or females over the age of 18 at the time of informed consent
* Access to a laptop, smartphone or tablet with a functioning microphone
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Fluency in English
* For depressed participant group: Current diagnosis of depression
* For non-depressed participant group: No current or prior diagnosis of depression

Exclusion Criteria:

* Visual impairment that would make it difficult for the participant to follow the instructions
* Motor impairment that would make it difficult for the participant to follow the instructions
* Any known history of neurodegenerative or Central Nervous System disorders (e.g. MS, Dementia, TBI, Stroke, etc.)
* Any known history of major psychiatric disorder other than depression (e.g. Bipolar Disorder, Schizophrenia, etc.)
* Any known history of substance abuse

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will enroll 225 men and women over the age of 18. 150 depressed participants will be recruited via an email from their treating psychiatrists. The researchers are collaborating with 2 psychiatric practices to recruit patients from.
  75 non-depressed participants will be recruited from the general population via Craigslist ads. Participants will go through a clinical evaluation with a mental health professional to rule out current episode of depression.
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2021-09-04 (Actual); Study Completion 2021-09-04 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of the Kintsugi's technology's prediction | July 30, 2021
  Sensitivity and specificity of the Kintsugi's technology's prediction compared to HAM-D and HAM-A scores.

SECONDARY OUTCOMES:
Sensitivity and specificity to depression at the PHQ-9 score of 10 | July 30, 2021
  Sensitivity and specificity of the Kintsugi's technology's prediction compared to PHQ-9 scores at a cutoff threshold of 10
Sensitivity and specificity to depression at the GAD-7 score of 10 | July 30, 2021
  Sensitivity and specificity of the Kintsugi's technology's prediction compared to GAD-7 scores at a cutoff threshold of 10

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - San Francisco Psychiatrists, Inc., San Francisco, California
  - Frontier Psychiatry, Billings, Montana